CLINICAL TRIAL: NCT03077958
Title: Total Knee Replacement With the Attune vs. the Press Fit Condylar (PFC) Sigma. Randomised Study of 50 Attune and 50 PFC Sigma Total Knee Replacements (TKRs)
Brief Title: Total Knee Replacement With the Attune vs. the Press Fit Condylar (PFC) Sigma.
Acronym: Att16SM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Karrholm, MD Professor in Orthopaedics, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Attune2016SM
Record Dates: First submitted 2016-04-28; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthrosis, Knee
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Patients with degenerative knee disease randomely receive one of two types of total knee prostheses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total Knee Replacement (2 different design) — Patients will randomely receive either Attune or PFC Sigma TKR
  Other Names: Attune or PFC Sigma TKR

SUMMARY:
100 knees with primary osteoarthritis and scheduled for a total knee replacement (TKR) will be recruited from our waiting list. The patients will be randomized to become operated with the Attune or PFC total knee arthroplasty. Randomisation will be done using envelopes. Patients can only participate with one knee.

DETAILED DESCRIPTION:
The Attune total knee replacement is a recently developed implant with the intention to improve the outcome after this procedure. One of the primary aims is to improve the kinematics of the knee in order to more closely mimic the normal knee. Thereby the patients are expected to experience improved function, better stability and less pain during activity. So far there are no randomized studies which have demonstrated this potential superior performance when compared to its predecessor, the PFC Sigma TKR. This study aims to evaluate the clinical outcome and the knee kinematics of the Attune knee using recognized clinical outcome parameters and dynamic radiostereometry. The PFC sigma knee will be used as control.

100 knees with primary osteoarthritis and scheduled for a total knee replacement (TKR) will be recruited from our waiting list. The patients will be randomized to become operated with the Attune or PFC total knee arthroplasty. Randomization will be done using envelopes. Patients can only participate with one knee.

Surgical procedure: The operations will be done according to our routines without use of bloodless field. Local analgesia will be infiltrated periarticulary during the operation. Cemented fixation will be used in all cases. So-called "fast-track"principles will be applied in both Groups.

Patients will be followed for five years.

ELIGIBILITY:
Patients with degenerative joint disease of the knee on our waiting list for a total knee replacement will be asked to participate in this study

Inclusion Criteria:

* Medial or lateral primary osteoarthritis (OA) Ahlbäck Grade 2-4
* Varus or valgus deformity ≤15 degrees, extension defect ≤15 degrees
* BMI <35
* ASA 1-3.
* Coming from independent living in own home
* Written informed consent

Exclusion Criteria:

* Cortisone treatment during the last 6 months before operation
* Neurological diseases with symptoms, stroke with sequel
* Endocrine diseases with symptoms
* OA secondary to trauma, infection, inflammatory disease or congenital and acquired deformities
* BMI >=35
* OA of the hip with symptoms. (Patients operated with total hip arthroplasty are accepted)
* Ongoing infection
* Unable or unwilling to participate in the follow-up.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-18 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | Preoperatively to 2 years
  The Oxford Knee Score (OKS) is a 12-item patient-reported outcome measure (PROM) specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is short, reproducible, valid and sensitive to clinically important changes.

SECONDARY OUTCOMES:
Patient satisfaction is reported on a visual analogue scale (VAS) 1-10 | Preoperatively to 2 years
  Patient satisfaction is reported on a visual analogue scale (VAS) 1-10
Knee Kinematics, (anterior-posterior translations and axial rotations) | 2 years
  Dynamic radiostereometric analysis with detailed recordings of the threedimensional motions of the knee during a step-up
Pain (VAS) | Preoperatively to 2 years
  Patient pain reported on Visual Analogue Scales(VAS) 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Johan Kärrholm, MD PhD Professor, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of Orthopaedics, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared with the sponsor (DePuy).